CLINICAL TRIAL: NCT01903915
Title: Resting-state Magnetic Resonance Imaging of Brain in Patients With Schizophrenia Compared With Healthy Controls to Prove the Association Between Social Cognition Dysfunction and Abnormality of Brain Function
Brief Title: Social Dysfunction and Brain Dysfunction in Patients With Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Sun Lee, Associate Professor, Department of Psychiatry, Asan Medical Center
Other Study IDs: 07052012
Record Dates: First submitted 2013-07-10; First posted 2013-07-19 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Schizophrenia; Social Cognition
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients: Schizophrenia group
- Control: Healthy control group

SUMMARY:
There were a few studies about the relationship of structural or functional abnormalities of brain and social cognitive dysfunctions in patients with schizophrenia. In addition, default network, which increases activity during mental explorations referenced to oneself including remembering, considering hypothetical social interactions, and thinking about one's own future, may be associated with social cognitive dysfunctions in patients with schizophrenia. Therefore, we will investigate the dysfunction of default network in patients with schizophrenia compared with healthy controls and the effect of default network dysfunctions on the social cognition in patients with schizophrenia.

ELIGIBILITY:
Patients group inclusion criteria:

* Right-handed
* Intelligent Quotient(IQ) above 80
* can read and understand the informed consent
* schizophrenia patients who was diagnosed from Structured Clinical Interview for Diagnostical and Statistical Manual of Mental Disorder 4th edition(DSM-IV, nonpatient version(SCID-NP) scales
* patient who has had reality distortion symptoms (like delusion or hallucination) in 5 years

Control group inclusion criteria :

* Right-handed
* IQ above 80
* do not have any diagnosis from SCID-NP scales
* do not have any family members who have psychiatric disorder

Exclusion criteria:

* have Illness which can affect brain structures and functions
* can't be taken magnetic resonance imaging(MRI)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients groups will be selected from psychiatric clinic in general hospital - Asan Medical Center.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-12 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Comparison of resting state functional MRI between schizophrenia patients and healthy controls | Baseline
  After subjects are enrolled the study, functional MRI of the brain will be measured on rest. They will lie down in MRI machine and just open their eyes. There is no tasks for functional MRI.
  Unless the subject don't have any contraindication for MRI, they can be take MRI of brain safely.
  Resting-state functional brain MRI Data from subjects will be analysed statistically. We will use programs for image processing and statistical work, such as REST, Statistical Parametric Mapping(SPM), Freesurfer. For comparison between two groups, student t-test will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Sun Lee, MD, Principal Investigator — Department of Psychiatry, Asan Medical Center
Locations (1):
- Department of psychiatry, Asan Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Garrity AG, Pearlson GD, McKiernan K, Lloyd D, Kiehl KA, Calhoun VD. Aberrant "default mode" functional connectivity in schizophrenia. Am J Psychiatry. 2007 Mar;164(3):450-7. doi: 10.1176/ajp.2007.164.3.450. PMID 17329470
- [Background] Hans S, Vaissiere J, Crevier-Buchman L, Laccourreye O, Brasnu D. Aerodynamic and acoustic parameters in CO2 laser posterior transverse cordotomy for bilateral vocal fold paralysis. Acta Otolaryngol. 2000 Mar;120(2):330-5. doi: 10.1080/000164800750001206. PMID 11603801
- [Background] Amodio DM, Kubota JT, Harmon-Jones E, Devine PG. Alternative mechanisms for regulating racial responses according to internal vs external cues. Soc Cogn Affect Neurosci. 2006 Jun;1(1):26-36. doi: 10.1093/scan/nsl002. PMID 18985098
- [Background] Newton DE, Thornton C, Konieczko KM, Jordan C, Webster NR, Luff NP, Frith CD, Dore CJ. Auditory evoked response and awareness: a study in volunteers at sub-MAC concentrations of isoflurane. Br J Anaesth. 1992 Aug;69(2):122-9. doi: 10.1093/bja/69.2.122. PMID 1389813
- [Background] Klee EW, Finlay JA, McDonald C, Attewell JR, Hebrink D, Dyer R, Love B, Vasmatzis G, Li TM, Beechem JM, Klee GG. Bioinformatics methods for prioritizing serum biomarker candidates. Clin Chem. 2006 Nov;52(11):2162-4. doi: 10.1373/clinchem.2006.072868. No abstract available. PMID 18061989
- [Background] Tan HY, Chen Q, Goldberg TE, Mattay VS, Meyer-Lindenberg A, Weinberger DR, Callicott JH. Catechol-O-methyltransferase Val158Met modulation of prefrontal-parietal-striatal brain systems during arithmetic and temporal transformations in working memory. J Neurosci. 2007 Dec 5;27(49):13393-401. doi: 10.1523/JNEUROSCI.4041-07.2007. PMID 18057197
- [Background] Keefe RS. Cognitive deficits in patients with schizophrenia: effects and treatment. J Clin Psychiatry. 2007;68 Suppl 14:8-13. PMID 18284272
- [Background] Fox MD, Snyder AZ, Zacks JM, Raichle ME. Coherent spontaneous activity accounts for trial-to-trial variability in human evoked brain responses. Nat Neurosci. 2006 Jan;9(1):23-5. doi: 10.1038/nn1616. Epub 2005 Dec 11. PMID 16341210
- [Background] Bogialli S, Curini R, Di Corcia A, Nazzari M, Sergi M. Confirmatory analysis of sulfonamide antibacterials in bovine liver and kidney: extraction with hot water and liquid chromatography coupled to a single- or triple-quadrupole mass spectrometer. Rapid Commun Mass Spectrom. 2003;17(11):1146-56. doi: 10.1002/rcm.1031. PMID 12772270
- [Background] Rieger JW, Kim A, Argyelan M, Farber M, Glazman S, Liebeskind M, Meyer T, Bodis-Wollner I. Cortical functional anatomy of voluntary saccades in Parkinson disease. Clin EEG Neurosci. 2008 Oct;39(4):169-74. doi: 10.1177/155005940803900404. PMID 19044213
- [Background] Barros M, Dempster EL, Illott N, Chabrawi S, Maior RS, Tomaz C, Silva MA, Huston JP, Mill J, Muller CP. Decreased methylation of the NK3 receptor coding gene (TACR3) after cocaine-induced place preference in marmoset monkeys. Addict Biol. 2013 May;18(3):452-4. doi: 10.1111/j.1369-1600.2011.00409.x. Epub 2011 Nov 9. PMID 22070124